CLINICAL TRIAL: NCT06203405
Title: The Efficacy of P0.1-guided Sedation Protocol in Critically Ill Patients Receiving Invasive Mechanical Ventilation: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Natdanai Ketdao, Principal Investigator, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI915/2023
Record Dates: First submitted 2023-12-07; First posted 2024-01-12 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Failure; Critical Illness; Respiratory Distress Syndrome, Adult; Lung Injury; Mechanical Ventilation Complication
Keywords: acute respiratory failure; sedation; respiratory drive monitoring; mechanical ventilation; intensive care unit
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness; Respiratory Distress Syndrome; Lung Injury | interventions — Fentanyl; Midazolam; Propofol; Dexmedetomidine; cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Titrating sedation targeting both optimal P0.1 and appropriate arousal level (Experimental): • Sedative drug adjustment to achieve the target of light sedation (RASS 0 to -2) and optimal respiratory drive measured by P0.1 of 1.5 - 3.5 cmH2O
  Interventions: Procedure: Titrating sedation targeting both optimal P0.1 and appropriate arousal level; Drug: Fentanyl; Drug: Midazolam; Drug: Propofol; Drug: Dexmedetomidine; Drug: Cisatracurium
- Titrating sedation targeting appropriate arousal level alone (No Intervention): • Sedative drug adjustment to achieve the target of light sedation (RASS 0 to -2) according to the standard clinical practice guidelines for managing pain and agitation for patients receiving mechanical ventilation in the ICU.

INTERVENTIONS:
Procedure: Titrating sedation targeting both optimal P0.1 and appropriate arousal level — * Sedation will be adjusted initially to target light sedation (RASS 0 to -2).
  * Sedative drugs include IV fentanyl (25-75 mcg/h), midazolam (0.02- 0.1 mg/kg/h), propofol (5-50 mcg/kg/min), dexmedetomidine (0.2-0.7 mcg/kg/h).
  * Deep sedation and neuromuscular blocking agents are allowed to facilitate mechanical ventilation adjustment in patients with refractory hypoxemia.
  * Dose of cisatracurium is 0.15-0.2 mg/kg intravenous bolus, then continuous infusion at 5 -20 mg/h.
  * Then sedation adjustment will be guided by P0.1 measurement.
  * If P0.1 value of 1.5-3.5 cmH2O is achieved, no further adjustment is required.
  * If P0.1 value <1.5, sedation will be reduced.
  * If P0.1 value >3.5, sedation will be increased.
  * If P0.1 value is still >3.5 with deep sedation, cisatracurium will be allowed and titrated until P0.1 value <3.5 cmH2O.
  * The study protocol will be continued for 48 hours or until the patients are considered ready for weaning.
  Arms: Titrating sedation targeting both optimal P0.1 and appropriate arousal level
Drug: Fentanyl — Continuous intravenous infusion of fentanyl 25-75 micrograms/hour
  Arms: Titrating sedation targeting both optimal P0.1 and appropriate arousal level
Drug: Midazolam — Continuous intravenous infusion of midazolam 0.02 - 0.1 milligrams/kilogram/hour
  Arms: Titrating sedation targeting both optimal P0.1 and appropriate arousal level
Drug: Propofol — Continuous intravenous infusion of propofol 5 - 50 micrograms/kilogram/minute
  Arms: Titrating sedation targeting both optimal P0.1 and appropriate arousal level
Drug: Dexmedetomidine — Continuous intravenous infusion of dexmedetomidine 0.2 - 0.7 micrograms/kilogram/hour
  Arms: Titrating sedation targeting both optimal P0.1 and appropriate arousal level
Drug: Cisatracurium — Continuous intravenous infusion of cisatracurium 5 - 20 milligrams/hour
  Arms: Titrating sedation targeting both optimal P0.1 and appropriate arousal level

SUMMARY:
This clinical trial aims to assess the efficacy of sedation protocol targeting optimal respiratory drive using P0.1 and arousal level compared with conventional sedation strategy (targeting arousal level alone) in patients requiring mechanical ventilation in the medical intensive care unit.

DETAILED DESCRIPTION:
Objective: to assess the efficacy of sedation protocol targeting optimal respiratory drive using P0.1 and RASS score compared with conventional sedation strategy (targeting RASS score alone) in patients requiring mechanical ventilation in the medical intensive care unit

The main questions it aims to answer are:

• Will titration of sedation targeting optimal respiratory drive assessed by P0.1 and arousal level improve outcomes in patients requiring mechanical ventilation in the medical ICU?

Study protocol Mechanically ventilated patients admitted to the medical ICU will be screened daily by the investigators. If the patients meet the eligibility criteria, they will be informed about the study protocol and potential risks and undergo informed consent. Then patients will be randomized in a 1:1 ratio and allocated to each study group (intervention and control group).

* After allocation, patients will be monitored for arousal level using RASS score and respiratory drive by P0.1 measured automatically from mechanical ventilators during the study period.
* Sedation and neuromuscular blocking agents used will be adjusted according to the group to which patients are allocated.
* Intervention group: Adjustment of sedation and neuromuscular blocking agents to achieve the target of light sedation (RASS 0 to -2) and optimal P0.1 (1.5 to 3.5 cmH2O) for 48 hours
* Control group: Adjustment of sedation to achieve the target of light sedation (RASS 0 to -2) alone for 48 hours

Researchers will compare the outcomes (rate of successful extubation, ICU and hospital mortality, ICU and hospital length of stay, duration of mechanical ventilation, amount and duration of sedation used during the study period) between the above sedation protocol (interventional group) and conventional sedation strategy (control group)

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the medical intensive care unit at Department of Medicine, Siriraj Hospital
2. Age ≥18 years old
3. Receiving mechanical ventilation due to acute respiratory failure within 72 hours before enrollment (including patients receiving mechanical ventilation before ICU admission)

Exclusion Criteria:

1. Patients receiving mechanical ventilation due to indications other than acute respiratory failure, such as postoperative procedures or airway protection in comatose patients
2. Patients receiving mechanical ventilation for >72 hours before enrollment
3. Patients receiving neuromuscular blocking agents prior to randomization
4. Patients with impaired secretion clearance or upper airway obstruction anticipating a tracheostomy
5. Patients with severe metabolic acidosis (arterial pH <7.2) who do not have a plan for renal replacement therapy
6. Patients intubated for neurological conditions, including intracranial hypertension, intracranial hemorrhage, large cerebral infarction, status epilepticus, or neuromuscular diseases
7. Post-cardiac arrest patients
8. Patients with severe liver dysfunction, including acute fulminant liver failure or cirrhosis with the Child-Pugh score B or C
9. Patients who have a previous allergy to any of the opioid, sedation, or neuromuscular blocking drugs
10. Pregnancy
11. Patients with do-not-resuscitate (DNR) orders or decisions to withhold life-sustaining treatments
12. Patients who refuse to participate in the study or cannot identify legally authorized representatives (LAR) within 24 hours after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful extubation within 14 days after randomization | 14 days after randomization
  Successful extubation within 14 days without reintubation within 28 days after ICU admission

SECONDARY OUTCOMES:
Successful extubation within 7 days after randomization | 7 days after randomization
  Successful extubation within 7 days without reintubation within 28 days after ICU admission
Successful extubation within 28 days after randomization | 28 days after randomization
  Successful extubation without reintubation within 28 days after ICU admission
Duration of mechanical ventilation | From date of intubation until the date of last successful extubation or date of death from any cause, whichever came first, assessed up to 28 days
  Time from intubation to the last successful extubation
Ventilator-free days to day 28 after randomization | 28 days after randomization
  Number of days alive without mechanical ventilation
Reintubation rate at 7 days after randomization | 7 days after randomization
  Number of reintubation within 7 days after randomization
Self extubation rate at 7 days after extubation | 7 days after randomization
  Number of self extubation (accidentally extubation without physician's order) within 7 days after randomization
Post-extubation respiratory failure | From date of randomization until the date of the first event of post-extubation respiratory failure or date of death from any cause or ICU discharge, whichever came first, assessed up to 28 days
  Patients who meet at least one of the following criteria within 72 hours after extubation: respiratory rate more than 35 breaths/minute, oxygen saturation less than 90% or PaO2 less than 80 mmHg despite receiving FiO2 >50%, respiratory acidosis with pH <7.35 or PaCO2 >50 mmHg or increase of 20% from baseline.
Tracheostomy | From date of randomization until the date of tracheostomy or date of death from any cause or ICU discharge, whichever came first, assessed up to 28 days
  Number of tracheostomy performed
Lung injury score on day 3 after randomization | 3 days after randomization
  Lung injury score on day 3 after randomization
Lung injury score on day 7 after randomization | 7 days after randomization
  Lung injury score on day 7 after randomization
PaO2/FiO2 ratio on day 3 after randomization | 3 days after randomization
  PaO2/FiO2 ratio on day 3 after randomization
PaO2/FiO2 ratio on day 7 after randomization | 7 days after randomization
  PaO2/FiO2 ratio on day 7 after randomization
Rates of new diagnosis of ARDS according to the new Berlin criteria after randomization | From date of randomization until the date of new onset ARDS diagnosis after randomization or date of death from any cause or ICU discharge, whichever came first, assessed up to 28 days
  Number of ARDS diagnoses after randomization
Delirium during ICU admission | From date of randomization until the date of diagnosis of delirium diagnosis or date of death from any cause or ICU discharge, whichever came first, assessed up to 28 days
  Delirium assessed by positive CAM-ICU criteria during ICU admission
Glasgow Outcome Scale (GOS) at hospital discharge | From date of randomization until the date of hospital discharge or date of death from any cause , whichever came first, assessed up to 28 days
  Functional status assessed by Glasgow Outcome Scale (GOS) at hospital discharge
  * Unabbreviated title: Glasgow Outcome Scale
  * Maximum score: 5 = good recovery
  * 4 = Moderate disability, 3 = Severe disability, 2 = Vegetative state
  * Minimum score: 1 = death (Higher scores mean better outcome)
ICU all-cause mortality | From date of randomization until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 28 days
  All-cause mortality during ICU admission
Hospital all-cause mortality | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 28 days
  All-cause mortality during hospital admission
28-day mortality after randomization | 28 days after randomization
  All-cause mortality during 28-day after randomization
ICU length of stay | From date of randomization until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 28 days
  Time from ICU admission to ICU discharge
Hospital length of stay | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 28 days
  Time from hospital admission to hospital discharge
Maximum infusion dose (per hour) of sedation | From date of sedation initiation until the date of sedation discontinuation or date of death from any cause, whichever came first, assessed up to 28 days
  Maximum infusion dose (per hour) of sedation used during the study period
Duration (days) of sedation | From date of sedation initiation until the date of sedation discontinuation or date of death from any cause, whichever came first, assessed up to 28 days
  Duration (days) of sedation used during the study period
Ventilator-associated pneumonia | From date of randomization until the date of first diagnosed ventilator-associated pneumonia or date of death from any cause, whichever came first, assessed up to 28 days
  Number of ventilator-associated pneumonia diagnosed after randomization
Barotrauma | From date of randomization until the date of first documented barotrauma or date of death from any cause, whichever came first, assessed up to 28 days
  Number of barotrauma (pneumothorax, pneumomediastinum, subcutaneous emphysema) occurred after randomization
Serious adverse events | From date of randomization until the date of first documented serious adverse events or date of death from any cause, whichever came first, assessed up to 28 days
  Number of serious adverse events (severe allergic reaction or anaphylaxis and propofol infusion syndrome defined as severe lactic acidosis and hypertriglyceridemia) occurred after randomization
Cardiac arrhythmia | From date of randomization until the date of first documented cardiac arrhythmia events or date of death from any cause, whichever came first, assessed up to 28 days
  Number of cardiac arrhythmia events occurred after randomization
Maximum infusion dose (per hour) of vasopressor | From date of vasopressor initiation until the date of vasopressor discontinuation or date of death from any cause, whichever came first, assessed up to 28 days
  Maximum infusion dose (per hour) of vasopressor used during the study period
Duration (days) of vasopressor | From date of vasopressor initiation until the date of vasopressor discontinuation or date of death from any cause, whichever came first, assessed up to 28 days
  Duration (days) of vasopressor used during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Tanuwong Viarasilpa, MD, Principal Investigator — Division of Critical Care, Department of Medicine, Siriraj Hospital, Mahidol University; Natdanai Ketdao, MD, Principal Investigator — Division of Critical Care, Department of Medicine, Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication of this study (after deidentification)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All IPD will become available starting briefly following a publication of the study with no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by institutional review board or ethical committee.

REFERENCES:
- [Background] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Background] Sklienka P, Frelich M, Bursa F. Patient Self-Inflicted Lung Injury-A Narrative Review of Pathophysiology, Early Recognition, and Management Options. J Pers Med. 2023 Mar 28;13(4):593. doi: 10.3390/jpm13040593. PMID 37108979
- [Background] Carteaux G, Parfait M, Combet M, Haudebourg AF, Tuffet S, Mekontso Dessap A. Patient-Self Inflicted Lung Injury: A Practical Review. J Clin Med. 2021 Jun 21;10(12):2738. doi: 10.3390/jcm10122738. PMID 34205783
- [Background] Spinelli E, Mauri T, Beitler JR, Pesenti A, Brodie D. Respiratory drive in the acute respiratory distress syndrome: pathophysiology, monitoring, and therapeutic interventions. Intensive Care Med. 2020 Apr;46(4):606-618. doi: 10.1007/s00134-020-05942-6. Epub 2020 Feb 3. PMID 32016537
- [Background] Spinelli E, Pesenti A, Slobod D, Fornari C, Fumagalli R, Grasselli G, Volta CA, Foti G, Navalesi P, Knafelj R, Pelosi P, Mancebo J, Brochard L, Mauri T. Clinical risk factors for increased respiratory drive in intubated hypoxemic patients. Crit Care. 2023 Apr 11;27(1):138. doi: 10.1186/s13054-023-04402-z. PMID 37041553
- [Background] Chanques G, Constantin JM, Devlin JW, Ely EW, Fraser GL, Gelinas C, Girard TD, Guerin C, Jabaudon M, Jaber S, Mehta S, Langer T, Murray MJ, Pandharipande P, Patel B, Payen JF, Puntillo K, Rochwerg B, Shehabi Y, Strom T, Olsen HT, Kress JP. Analgesia and sedation in patients with ARDS. Intensive Care Med. 2020 Dec;46(12):2342-2356. doi: 10.1007/s00134-020-06307-9. Epub 2020 Nov 10. PMID 33170331
- [Background] Goligher EC, Jonkman AH, Dianti J, Vaporidi K, Beitler JR, Patel BK, Yoshida T, Jaber S, Dres M, Mauri T, Bellani G, Demoule A, Brochard L, Heunks L. Clinical strategies for implementing lung and diaphragm-protective ventilation: avoiding insufficient and excessive effort. Intensive Care Med. 2020 Dec;46(12):2314-2326. doi: 10.1007/s00134-020-06288-9. Epub 2020 Nov 2. PMID 33140181
- [Background] Dzierba AL, Khalil AM, Derry KL, Madahar P, Beitler JR. Discordance Between Respiratory Drive and Sedation Depth in Critically Ill Patients Receiving Mechanical Ventilation. Crit Care Med. 2021 Dec 1;49(12):2090-2101. doi: 10.1097/CCM.0000000000005113. PMID 34115638
- [Background] Wongtangman K, Grabitz SD, Hammer M, Wachtendorf LJ, Xu X, Schaefer MS, Fassbender P, Santer P, Kassis EB, Talmor D, Eikermann M; SICU Optimal Mobilization Team (SOMT) Group. Optimal Sedation in Patients Who Receive Neuromuscular Blocking Agent Infusions for Treatment of Acute Respiratory Distress Syndrome-A Retrospective Cohort Study From a New England Health Care Network. Crit Care Med. 2021 Jul 1;49(7):1137-1148. doi: 10.1097/CCM.0000000000004951. PMID 33710031
- [Background] Jackson DL, Proudfoot CW, Cann KF, Walsh TS. The incidence of sub-optimal sedation in the ICU: a systematic review. Crit Care. 2009;13(6):R204. doi: 10.1186/cc8212. Epub 2009 Dec 16. PMID 20015357
- [Background] Kassis EB, Beitler JR, Talmor D. Lung-protective sedation: moving toward a new paradigm of precision sedation. Intensive Care Med. 2023 Jan;49(1):91-94. doi: 10.1007/s00134-022-06901-z. Epub 2022 Oct 14. No abstract available. PMID 36239747
- [Background] Bertoni M, Spadaro S, Goligher EC. Monitoring Patient Respiratory Effort During Mechanical Ventilation: Lung and Diaphragm-Protective Ventilation. Crit Care. 2020 Mar 24;24(1):106. doi: 10.1186/s13054-020-2777-y. PMID 32204729
- [Background] Rittayamai N, Beloncle F, Goligher EC, Chen L, Mancebo J, Richard JM, Brochard L. Effect of inspiratory synchronization during pressure-controlled ventilation on lung distension and inspiratory effort. Ann Intensive Care. 2017 Oct 6;7(1):100. doi: 10.1186/s13613-017-0324-z. PMID 28986852
- [Background] Telias I, Junhasavasdikul D, Rittayamai N, Piquilloud L, Chen L, Ferguson ND, Goligher EC, Brochard L. Airway Occlusion Pressure As an Estimate of Respiratory Drive and Inspiratory Effort during Assisted Ventilation. Am J Respir Crit Care Med. 2020 May 1;201(9):1086-1098. doi: 10.1164/rccm.201907-1425OC. PMID 32097569
- [Background] Beloncle F, Piquilloud L, Olivier PY, Vuillermoz A, Yvin E, Mercat A, Richard JC. Accuracy of P0.1 measurements performed by ICU ventilators: a bench study. Ann Intensive Care. 2019 Sep 13;9(1):104. doi: 10.1186/s13613-019-0576-x. PMID 31520230
- [Background] de Vries HJ, Tuinman PR, Jonkman AH, Liu L, Qiu H, Girbes ARJ, Zhang Y, de Man AME, de Grooth HJ, Heunks L. Performance of Noninvasive Airway Occlusion Maneuvers to Assess Lung Stress and Diaphragm Effort in Mechanically Ventilated Critically Ill Patients. Anesthesiology. 2023 Mar 1;138(3):274-288. doi: 10.1097/ALN.0000000000004467. PMID 36520507
- [Background] Writing Group for the PReVENT Investigators; Simonis FD, Serpa Neto A, Binnekade JM, Braber A, Bruin KCM, Determann RM, Goekoop GJ, Heidt J, Horn J, Innemee G, de Jonge E, Juffermans NP, Spronk PE, Steuten LM, Tuinman PR, de Wilde RBP, Vriends M, Gama de Abreu M, Pelosi P, Schultz MJ. Effect of a Low vs Intermediate Tidal Volume Strategy on Ventilator-Free Days in Intensive Care Unit Patients Without ARDS: A Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1872-1880. doi: 10.1001/jama.2018.14280. PMID 30357256
- [Background] Grasselli G, Calfee CS, Camporota L, Poole D, Amato MBP, Antonelli M, Arabi YM, Baroncelli F, Beitler JR, Bellani G, Bellingan G, Blackwood B, Bos LDJ, Brochard L, Brodie D, Burns KEA, Combes A, D'Arrigo S, De Backer D, Demoule A, Einav S, Fan E, Ferguson ND, Frat JP, Gattinoni L, Guerin C, Herridge MS, Hodgson C, Hough CL, Jaber S, Juffermans NP, Karagiannidis C, Kesecioglu J, Kwizera A, Laffey JG, Mancebo J, Matthay MA, McAuley DF, Mercat A, Meyer NJ, Moss M, Munshi L, Myatra SN, Ng Gong M, Papazian L, Patel BK, Pellegrini M, Perner A, Pesenti A, Piquilloud L, Qiu H, Ranieri MV, Riviello E, Slutsky AS, Stapleton RD, Summers C, Thompson TB, Valente Barbas CS, Villar J, Ware LB, Weiss B, Zampieri FG, Azoulay E, Cecconi M; European Society of Intensive Care Medicine Taskforce on ARDS. ESICM guidelines on acute respiratory distress syndrome: definition, phenotyping and respiratory support strategies. Intensive Care Med. 2023 Jul;49(7):727-759. doi: 10.1007/s00134-023-07050-7. Epub 2023 Jun 16. PMID 37326646
- [Background] Brenner M, Mukai DS, Russell JE, Spiritus EM, Wilson AF. A new method for measurement of airway occlusion pressure. Chest. 1990 Aug;98(2):421-7. doi: 10.1378/chest.98.2.421. PMID 2376174
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Seo Y, Lee HJ, Ha EJ, Ha TS. 2021 KSCCM clinical practice guidelines for pain, agitation, delirium, immobility, and sleep disturbance in the intensive care unit. Acute Crit Care. 2022 Feb;37(1):1-25. doi: 10.4266/acc.2022.00094. Epub 2022 Feb 28. PMID 35279975
- [Background] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Moss M, Huang DT, Brower RG, Ferguson ND, Ginde AA, Gong MN, Grissom CK, Gundel S, Hayden D, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Khan A, Liu KD, Talmor D, Thompson BT, Ulysse CA, Yealy DM, Angus DC. Early Neuromuscular Blockade in the Acute Respiratory Distress Syndrome. N Engl J Med. 2019 May 23;380(21):1997-2008. doi: 10.1056/NEJMoa1901686. Epub 2019 May 19. PMID 31112383
- [Background] Marra A, Ely EW, Pandharipande PP, Patel MB. The ABCDEF Bundle in Critical Care. Crit Care Clin. 2017 Apr;33(2):225-243. doi: 10.1016/j.ccc.2016.12.005. PMID 28284292
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Tongyoo S, Tantibundit P, Daorattanachai K, Viarasilpa T, Permpikul C, Udompanturak S. High-flow nasal oxygen cannula vs. noninvasive mechanical ventilation to prevent reintubation in sepsis: a randomized controlled trial. Ann Intensive Care. 2021 Sep 14;11(1):135. doi: 10.1186/s13613-021-00922-5. PMID 34523035
- [Background] Sandhu RS, Pasquale MD, Miller K, Wasser TE. Measurement of endotracheal tube cuff leak to predict postextubation stridor and need for reintubation. J Am Coll Surg. 2000 Jun;190(6):682-7. doi: 10.1016/s1072-7515(00)00269-6. PMID 10873003
- [Background] Cheng KC, Hou CC, Huang HC, Lin SC, Zhang H. Intravenous injection of methylprednisolone reduces the incidence of postextubation stridor in intensive care unit patients. Crit Care Med. 2006 May;34(5):1345-50. doi: 10.1097/01.CCM.0000214678.92134.BD. PMID 16540947
- [Background] Fan T, Wang G, Mao B, Xiong Z, Zhang Y, Liu X, Wang L, Yang S. Prophylactic administration of parenteral steroids for preventing airway complications after extubation in adults: meta-analysis of randomised placebo controlled trials. BMJ. 2008 Oct 20;337:a1841. doi: 10.1136/bmj.a1841. PMID 18936064
- [Background] Pluijms WA, van Mook WN, Wittekamp BH, Bergmans DC. Postextubation laryngeal edema and stridor resulting in respiratory failure in critically ill adult patients: updated review. Crit Care. 2015 Sep 23;19(1):295. doi: 10.1186/s13054-015-1018-2. PMID 26395175
- [Background] Lee CH, Peng MJ, Wu CL. Dexamethasone to prevent postextubation airway obstruction in adults: a prospective, randomized, double-blind, placebo-controlled study. Crit Care. 2007;11(4):R72. doi: 10.1186/cc5957. PMID 17605780
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357
- [Background] Klompas M, Branson R, Cawcutt K, Crist M, Eichenwald EC, Greene LR, Lee G, Maragakis LL, Powell K, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia, ventilator-associated events, and nonventilator hospital-acquired pneumonia in acute-care hospitals: 2022 Update. Infect Control Hosp Epidemiol. 2022 Jun;43(6):687-713. doi: 10.1017/ice.2022.88. Epub 2022 May 20. PMID 35589091
- [Background] Singh A, Anjankar AP. Propofol-Related Infusion Syndrome: A Clinical Review. Cureus. 2022 Oct 17;14(10):e30383. doi: 10.7759/cureus.30383. eCollection 2022 Oct. PMID 36407194
- [Background] Murray JF, Matthay MA, Luce JM, Flick MR. An expanded definition of the adult respiratory distress syndrome. Am Rev Respir Dis. 1988 Sep;138(3):720-3. doi: 10.1164/ajrccm/138.3.720. No abstract available. PMID 3202424
- [Background] Matthay MA, Arabi Y, Arroliga AC, Bernard G, Bersten AD, Brochard LJ, Calfee CS, Combes A, Daniel BM, Ferguson ND, Gong MN, Gotts JE, Herridge MS, Laffey JG, Liu KD, Machado FR, Martin TR, McAuley DF, Mercat A, Moss M, Mularski RA, Pesenti A, Qiu H, Ramakrishnan N, Ranieri VM, Riviello ED, Rubin E, Slutsky AS, Thompson BT, Twagirumugabe T, Ware LB, Wick KD. A New Global Definition of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2024 Jan 1;209(1):37-47. doi: 10.1164/rccm.202303-0558WS. PMID 37487152